CLINICAL TRIAL: NCT00027534
Title: A Phase I Study Of Active Immunotherapy With Autologous Dendritic Cells Infected With CEA-6D Expressing Fowlpox -Tricom In Patients With Advanced Or Metastatic Malignancies Expressing CEA
Brief Title: Vaccine Therapy in Treating Patients With Advanced or Metastatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Michael Morse, MD (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Michael Morse, MD, Principal Investigator, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2840; 1R21CA094523 (NIH); 2840 (Other: Duke IRB); CDR0000069041
Record Dates: First submitted 2001-12-07; First posted 2003-01-27 (Estimated); Last update posted 2014-09-08 (Estimated); Status verified 2014-09

CONDITIONS: Breast Cancer; Colorectal Cancer; Gallbladder Cancer; Gastric Cancer; Head and Neck Cancer; Liver Cancer; Ovarian Cancer; Pancreatic Cancer; Testicular Germ Cell Tumor
Keywords: recurrent colon cancer; stage III colon cancer; stage IV colon cancer; recurrent breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV breast cancer; recurrent gastric cancer; stage III gastric cancer; stage IV gastric cancer; recurrent pancreatic cancer; stage II pancreatic cancer; stage III pancreatic cancer; recurrent rectal cancer; stage III rectal cancer; stage IV rectal cancer; advanced adult primary liver cancer; recurrent adult primary liver cancer; recurrent gallbladder cancer; unresectable gallbladder cancer; thyroid gland medullary carcinoma; recurrent salivary gland cancer; stage III salivary gland cancer; stage IV salivary gland cancer; Paget disease of the breast with intraductal carcinoma; Paget disease of the breast with invasive ductal carcinoma; adult primary hepatocellular carcinoma; diffuse adenocarcinoma of the stomach; intestinal adenocarcinoma of the stomach; mixed adenocarcinoma of the stomach; adenocarcinoma of the colon; adenocarcinoma of the gallbladder; adenocarcinoma of the rectum; recurrent malignant testicular germ cell tumor; stage II malignant testicular germ cell tumor; stage III malignant testicular germ cell tumor; male breast cancer; adenocarcinoma of the pancreas; cholangiocarcinoma of the gallbladder; salivary gland adenocarcinoma; ovarian endometrioid adenocarcinoma; stage IV pancreatic cancer
MeSH Terms: conditions — Breast Neoplasms; Colorectal Neoplasms; Gallbladder Neoplasms; Stomach Neoplasms; Head and Neck Neoplasms; Liver Neoplasms; Ovarian Neoplasms; Pancreatic Neoplasms; Testicular Germ Cell Tumor; Colonic Neoplasms; Rectal Neoplasms; Carcinoma, Hepatocellular; Carcinoma, Medullary; Salivary Gland Neoplasms; Testicular Neoplasms; Breast Neoplasms, Male

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TRICOM-CEA(6D) (Experimental): Subjects receiving TRICOM-CEA(6D)
  Interventions: Biological: TRICOM-CEA(6D)

INTERVENTIONS:
Biological: TRICOM-CEA(6D) — dendritic cells loaded with TRICOM-CEA(6D)
  Other Names: recombinant fowlpox-CEA(6D)/TRICOM vaccine

SUMMARY:
RATIONALE: Vaccines made from a person's white blood cells that have been treated in the laboratory may make the body build an immune response to kill tumor cells.

PURPOSE: Phase I trial to study the effectiveness of vaccine therapy in treating patients who have advanced or metastatic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the safety and feasibility of active immunotherapy comprising autologous dendritic cells infected with recombinant fowlpox-CEA-TRICOM vaccine in patients with advanced or metastatic malignancies expressing CEA.
* Assess the CEA-specific immune response of patients treated with this regimen.
* Assess, in a preliminary manner, the clinical response rate of patients treated with this regimen.

OUTLINE: This is a dose-escalation study.

Autologous dendritic cells (ADCs) are harvested and infected with fowlpox-CEA-TRICOM vaccine. Patients receive the infected ADCs intradermally and subcutaneously (SC) followed by ADCs mixed with CMV pp65 peptide and ADCs mixed with tetanus toxoid SC and intradermally on day 1. Treatment repeats every 3 weeks for a total of 4, 8, or 12 immunizations in the absence of unacceptable toxicity.

Cohorts of 6 patients receive an escalating number of immunizations until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity.

Patients are followed every 3 months for 1 year.

PROJECTED ACCRUAL: A total of 6-18 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed advanced or metastatic malignancy expressing CEA

  * Metastatic disease meeting one of the following criteria:

    * Measurable or nonmeasurable
    * History of metastases but no current evidence of disease, meeting one of the following criteria:

      * Unresectable peritoneal or lymph node metastases that cannot be detected by imaging
      * Treated or resected metastatic disease considered at high risk of recurrence (predicted 5-year disease-free survival of less than 50%)

        * Must have completed treatment that rendered no evidence of disease within the past year
* CEA-expressing malignancy is defined by any of the following:

  * Immunohistochemical staining (at least 50% of the tumor has at least a moderate intensity of staining)
  * CEA level in peripheral blood greater than 2.5 µg/L
  * Tumor known to be universally CEA positive (e.g., colon and rectal cancer)
* Received prior therapy with possible survival benefit or refused such therapy
* Prior resection of brain metastases allowed provided no metastasis by CT scan or MRI of the brain within 1 month of enrollment
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age

* 18 and over Sex
* Male or female Menopausal status
* Not specified Performance status
* Karnofsky 70-100% Life expectancy
* More than 6 months

Hematopoietic

* WBC at least 3,000/mm^3
* Absolute lymphocyte count at least 1,000/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 9 g/dL (transfusion or epoetin alfa allowed) Hepatic
* Bilirubin less than 2.0 mg/dL
* SGOT/SGPT less than 1.5 times upper limit of normal
* No active acute or chronic viral hepatitis
* Hepatitis B surface antigen negative
* Hepatitis C negative
* No other hepatic disease that would preclude study entry

Renal

* Creatinine less than 2.5 mg/dL
* No active acute or chronic urinary tract infection

Cardiovascular

* No New York Heart Association class III or IV heart disease Immunologic
* HIV negative
* No history of autoimmune disease, including, but not limited to, the following:

  * Inflammatory bowel disease
  * Systemic lupus erythematosus
  * Rheumatoid arthritis
  * Ankylosing spondylitis
  * Scleroderma
  * Multiple sclerosis
* No allergy to eggs or any component of study vaccine Other
* No active acute or chronic infection
* No concurrent serious acute or chronic illness that would preclude study entry
* No other medical or psychological impediment that would preclude study entry
* No other malignancy within the past 5 years except nonmelanoma skin cancer, controlled carcinoma in situ of the cervix, or controlled superficial bladder cancer
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy

* At least 4 weeks since prior biologic therapy and recovered
* No other concurrent immunotherapy

Chemotherapy

* At least 4 weeks since prior chemotherapy and recovered
* No concurrent chemotherapy

Endocrine therapy

* At least 4 weeks since prior hormonal therapy and recovered
* At least 6 weeks since prior steroids except steroids used as premedication for chemotherapy or for contrast-enhanced studies
* No concurrent steroids

Radiotherapy

* Prior palliative radiotherapy (including systemic radiolabeled compounds) for unstable or painful bone metastases in weight-bearing bones may be allowed
* At least 4 weeks since prior radiotherapy and recovered
* No concurrent radiotherapy

Surgery

* Not specified

Other

* At least 4 weeks since any other prior therapy (including experimental therapy) and recovered
* No concurrent immunosuppressives (e.g., azathioprine or cyclosporine)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2002-01; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Safety | 12-36 weeks
  The primary objective of this protocol is to determine the safety and feasibility of rF-CEA(6D)-TRICOM loaded DC in, subjects with metastatic, CEA expressing malignancies.

SECONDARY OUTCOMES:
Immune response | 12-36 weeks
  The immune response to the injections of the TRICOM-CEA(6D) antigen loaded DC will be evaluated

CONTACTS AND LOCATIONS:
Overall Officials: Herbert K. Lyerly, MD, Study Chair — Duke Cancer Institute
Locations (1):
- Duke Comprehensive Cancer Center, Durham, North Carolina, United States